CLINICAL TRIAL: NCT05652855
Title: Phase 1/2, Two-Part, Multi-center, Open-label, Dose Escalation and Dose Expansion First-In-Human Study to Evaluate the Safety/Tolerability, Pharmacokinetics and Efficacy of MHB088C in Participants With Advanced or Metastatic Solid Tumors
Brief Title: Study of MHB088C in Participants With Advanced or Metastatic Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Minghui Pharmaceutical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHB088C-CP001EN
Record Dates: First submitted 2022-11-30; First posted 2022-12-15 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Intervention Model Description: Single group contains two study parts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MHB088C administered (Experimental): MHB088C will be administered intravenously at a frequency of once every 2 weeks (Q2W).
  Interventions: Drug: MHB088C for Injection

INTERVENTIONS:
Drug: MHB088C for Injection — MHB088C for Injection, an antibody drug-conjugated molecule (ADC)

SUMMARY:
This study will evaluate the safety/tolerability, pharmacokinetics and efficacy of MHB088C in participants with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This study is the first-in-human (FIH) trial of MHB088C, which contains two parts: dose escalation (part one) and dose expansion (part two).

Part one: Dose Escalation Study of MHB088C Monotherapy in Participants with Advanced or Metastatic Malignant Solid Tumors The dose escalation part is an open-label, multi-center study in which the eligible participants with advanced or metastatic solid tumors will be enrolled to receive MHB088C monotherapy to assess the safety and tolerability of MHB088C in participants with advanced or metastatic solid tumors, to determine the maximum tolerated dose (MTD) of MHB088C, and to assess its pharmacokinetic profile and preliminary efficacy.

The dose expansion part is an open-label, multi-center, multi-cohort expansion study in which participants with advanced or metastatic solid tumors of some predefined cancer types will be enrolled to receive MHB088C monotherapy. Participants with same types of solid tumors will be randomised into different selected dose groups and will be treated with the corresponding dose. This study is designed to assess the preliminary efficacy and safety of MHB088C monotherapy in participants with some types of advanced or metastatic solid tumors, so as to determine the recommended phase 2 dose (RP2D); and to assess the immunogenicity and pharmacokinetic profiles of MHB088C.

ELIGIBILITY:
Inclusion Criteria:

-

Participants enrolled must meet all of the following criteria:

General conditions

1. Participants voluntarily agree to participate in the study and sign the Informed Consent Form.
2. Aged ≥18years, without gender limitation.
3. Has an Eastern Cooperative Oncology Group Performance score (ECOG) 0 ~ 1.
4. Has a life expectancy of ≥ 3 months.
5. Eligible participants of childbearing potential (males and females) must agree to take highly reliable contraceptive measures (hormone or barrier method, or absolute abstinence, etc.) with their partners during the study and within at least 90 days after the last dose and agree not to retrieve, freeze or donate sperm or ova from screening to at least 3 months after the last dose of investigational drug; female participants of childbearing potential must have a negative results of blood pregnancy test within 7 days before the first dose of investigational drug, and must be non-lactating.
6. Understand study requirements, willing and able to comply with study and follow-up procedures.

   Neoplasm-related criteria
7. Part one: Histologically or cytologically confirmed unresectable advanced or metastatic malignant solid tumors, that is progressed or intolerant with standard of care (SOC), or for which no SOC regimens are available;
8. Part two: Histologically or cytologically confirmed unresectable advanced or metastatic malignant solid tumors, that is relapsed or progressed following systemic treatment or no standard of care is available, including but not limited to the following types: non-small cell lung cancer (NSCLC); small cell lung cancer (SCLC); esophageal squamous cell carcinoma (ESCC); castration-resistant prostate cancer (CRPC); melanoma (MEL); colorectal cancer (CRC); pancreatic ductal adenocarcinoma (PDAC); head and neck squamous cell carcinoma (HNSCC); hepatocellular carcinoma (HCC); ovarian cancer (OC); endometrial cancer (EC); thyroid cancer (TC); and sarcoma (SARC).

   1. Additional inclusion criteria for participants with NSCLC:

      Histologically or cytologically documented unresectable advanced or metastatic NSCLC and previous progressed during or after systematic treatment with platinum-contained doublet regimens chemotherapy and immune-checkpoint inhibitors (ICIs); refractory, intolerant or not suitable to the target therapy as per investigator discretion for participants with driver gene mutation.
   2. Additional inclusion criteria for participants with SCLC:

      Histologically or cytologically documented unresectable advanced or metastatic SCLC and previous progressed during or after ≥1 lines of systematic treatment with platinum-based, doublet regimens chemotherapy and ICIs.
   3. Additional inclusion criteria for participants with ESCC:

      Histologically or cytologically documented unresectable advanced or metastatic ESCC previous progressed during or after≥1 line platinum-based of systemic treatment.
   4. Additional inclusion criteria for participants with CRPC:

      Histologically or cytologically documented CRPC without neuroendocrine differentiation or small cell elements; Underwent surgical or medical castration, with testosterone levels below 50 ng/dL; Objective progression as determined by radiographic after androgen deprivation therapy; Relapsed or progressed during or after at least one of the following medicines: abiraterone, enzalutamide, apalutamide, or darolutamide; Relapsed or progressed during or after≥ 1 line of docetaxel/mitoxantrone-based cytotoxic chemotherapy regimens for metastatic CRPC; With at least 1 documented lesion confirmed by either a bone scan or a CT/MRI scan.
   5. Additional inclusion criteria for participants with MEL:

      Histologically or cytologically documented unresectable advanced or metastatic MEL and previous progressed during or after ≥1 line of systemic therapy including ICIs
   6. Additional inclusion criteria for participants with CRC:

      Histologically or cytologically documented unresectable advanced or metastatic CRC and previous progressed during or after systematic chemotherapy containing oxaliplatin, irinotecan, fluorouracil and immunotherapy (for participants with MSI-H/dMMR).
   7. Additional inclusion criteria for participants with PDAC:

      Histologically or cytologically documented unresectable advanced or metastatic PDAC and previous progressed during or after ≥ 1 line of systemic therapy in neoadjuvant, adjuvant, locally advanced or metastatic setting.
   8. Additional inclusion criteria for participants with HNSCC:

      Histologically or cytologically documented unresectable advanced or metastatic HNSCC and previous progressed during or after ≥ 1 line of systemic therapy, including platinum-based chemotherapy and ICIs (combined or sequential therapy).
   9. Additional inclusion criteria for participants with HCC:

      Histologically or cytologically documented unresectable advanced or metastatic HCC and previously progressed during or after ≥ 1 line of systemic therapy, including anti-vascular therapy and/or ICI therapy.
   10. Additional inclusion criteria for participants with OC:

       Histologically or cytologically documented unresectable advanced or metastatic OC including less-common histology per National Comprehensive Cancer Network (NCCN) of epithelial ovarian cancer as well as fallopian tube cancer and primary peritoneal cancer and have relapsed or progressed during or after ≥ 1 line of platinum-based systemic chemotherapy treatment.
   11. Additional inclusion criteria for participants with EC:

       Histologically or cytologically documented unresectable advanced or metastatic EC and recurrence after radical therapy, and previously treated and progressed during or after ≥ 1 line of standard systemic therapy.
   12. Additional inclusion criteria for participants with TC:

       Histologically or cytologically documented unresectable advanced or metastatic TC and previous progressed during or after ≥ 1 line of systemic therapy including platinum-based chemotherapy or targeted therapy.
   13. Additional inclusion criteria for participants with SARC:

   Histologically or cytologically documented unresectable advanced or metastatic SARC and previous progressed during or after ≥ 1 prior line of systemic therapy including doxorubicin-based chemotherapy.
9. Agree to provide the pre-existing diagnostic tumor samples for retrospective testing of target expression and other biomarkers (participants who agree but are unable to provide pre-existing tumor sample may also be enrolled). There is no minimum target expression level required for inclusion.
10. Has at least one measurable tumor lesion as per RECIST v1.1(generally, previously irradiated areas or locoregionally treated sites will not be considered as measurable lesions, unless these lesions have clearly progressed or still exist three months after radiotherapy); for participants with CRPC, evaluable lesions as defined by PCWG3 criteria or at least one measurable soft tissue tumor lesion as per RECIST v1.1 are required.

    Adequate bone marrow reserve and organ functions:
11. Adequate bone marrow reserve (without transfusion or colony-stimulating factor or equivalent within7 days before the screening period testing); Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L; Platelet count ≥ 100 × 10^9/L; Hemoglobin ≥ 9.0 g/dL.
12. Adequate hepatic function (with reference to normal values specified by the clinical study site):

    Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); TBIL ≤ 2 × ULN if Gilbert's syndrome is present; TBIL ≤ 3.0 × ULN is permitted if direct bilirubin (DBIL) suggests extrahepatic obstruction.

    Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) shall be ≤ 3 × ULN with non-hepatic tumors and without hepatic metastasis; AST and ALT shall be ≤ 5.0 × ULN with hepatic tumors or hepatic metastasis;
13. Adequate renal function (with reference to normal values specified by the clinical study site):

    Creatinine (Cr) ≤ 1.5 × ULN; when Cr > 1.5 × ULN, only participants with creatinine clearance (Ccr) ≥ 50 mL/min can be enrolled (using Cockcroft-Gault formula);
14. Adequate coagulation function:

    Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN, and international normalized ratio (INR) ≤ 1.5 × ULN.
15. Adequate cardiac function:

Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram within 28 days before enrollment; New York Heart Association (NYHA) Class < grade 3.

Exclusion Criteria:

-

Participants will be not enrolled if they meet any of the following exclusion criteria:

Neoplasm-related criteria:

1. Has more than 2 primary malignancies (except curatively treated non-melanoma skin cancer, in situ disease, and other curatively malignancies have considered cured) within 5 years before signing of Informed Consent Form.
2. Has received chemotherapy within 3 weeks, or have received anti-tumor treatment including radiation therapy, biologic therapy, endocrine therapy, immunotherapy, etc. within 4 weeks before the first dose of investigational product; or participants with the following conditions:

   Medication of nitrosourea or mitomycin C within 6 weeks before the first dose of investigational drug; Medication of oral fluoropyrimidines and small molecule targeted agents within 5 half-lives before the first dose of investigational drug; Medication of traditional Chinese medicine with anti-tumor indication within 2 weeks before the first dose of investigational drug.
3. Medication of other unmarketed investigational drugs or therapies within 4 weeks before the first dose of investigational drug.
4. Presence of brain metastases and/or leptomeningeal carcinomatosis. Participants previously treated for brain metastases may be considered to be enrolled in this study, provided they have been in stable condition for at least 1 month, have no progression confirmed by radiographic examination within 4 weeks before the first dose of study treatment, all neurological symptoms have stabled, there is no evidence of new or enlarging brain metastases, and radiation or surgical therapy is discontinued for at least 28 days before the first dose of study treatment and steroid therapy at the dose of ≤10 mg/day or similar drugs at equivalent dose within 14 days before the first dose and during the study. This exception does not include carcinomatous meningitis, which should be excluded regardless of clinical stability.
5. Has previously received same target therapy.
6. Has adverse reactions from previous anti-tumor treatment that have not recovered to ≤ CTCAE 5.0 Grade 1 (except for toxicities without safety risks as determined by the investigator, such as alopecia, hypothyroidism stably managed by hormone replacement therapy, etc.).

   General conditions:
7. Has underwent major organ surgery (excluding biopsy) or significant trauma within 4 weeks before the first dose of investigational drug or requiring elective surgery during the study.
8. Has vaccinated with attenuated live vaccines (except for SARS-CoV-2 vaccination) within 4 weeks before the first dose of investigational drug.
9. Has mucosal or internal bleeding for non-traumatic reason within 4 weeks before the first dose of investigational drug.
10. Has received treatment with systemic corticosteroids (prednisone at >10 mg/day, or similar drugs at equivalent dose) or other immunosuppressive agents within 14 days before the first dose of investigational drug, with the following exceptions:

    Treatment with topical, ocular, intra-articular, intranasal, and inhaled corticosteroids; Short-term use of glucocorticoids for prophylaxis (e.g., prevention of contrast media allergy).
11. Has pulmonary disease that severely impact pulmonary function, including, but not limited to, potential pulmonary disease, any autoimmune diseases, connective tissue diseases, or inflammatory diseases involving the pulmonary, or pneumonectomy.
12. Has history of non-infectious interstitial lung disease (ILD)/pneumonitis that required steroids, or current ILD/pneumonia, or suspected ILD/pneumonia that cannot be excluded by imaging examination at screening.
13. Has active pulmonary tuberculosis.
14. Has active infection requiring systemic therapy.
15. Has positive results in virus serology tests (participants receiving antiviral prophylaxis other than interferon are allowed to be enrolled):

    Positive result of HIV antibody; Or, positive for both HBsAg and HBV-DNA (i.e., HBV DNA ≥LLOD); Or, positive for HCV Ab (except HCV-RNA < LLOD).
16. Has positive result for covid-19 nucleic acid test.
17. Medical history of serious cardiovascular and cerebrovascular diseases, including but not limited to:

    Severe arrhythmia or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, or atrioventricular block Ⅱ~Ⅲ degree; Fridericia-corrected QT interval (QTcF) prolongation to >450 milisecond (ms) for males and > 470 ms for females; Acute coronary syndrome, aortic dissection, stroke or transient ischemic attack (TIA) within 6 months before the first dose; New myocardial infarction or unstable angina within 6 months before the first dost; Clinically uncontrolled hypertension;
18. Has clinically uncontrolled effusion in third spacing, deemed as inappropriate for enrollment by the investigator.
19. Hypersensitivity or delayed hypersensitivity to certain components or analogues of the investigational drug.
20. Has drug abuse or any other medical conditions, such as clinically significant psychological conditions that may interfere with study participation or the results of the clinical study as per investigator discretion.
21. Has alcohol or drug dependence.
22. Females who are pregnant or breastfeeding, or males/females who plan to father a child/get pregnant.
23. Poor compliance as per investigator discretion, has history of other serious systemic diseases, or unsuitable to participate this clinical study for some reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-01-23 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the incidence of adverse events (AEs) | through study completion, an average of 1 year
  Adverse events was assessed by investigator(s) according to NCI-CTCAE v5.0
Evaluate the incidence of dose-limiting toxicities (DLTs) | through study completion, an average of 1 year
  Dose-limiting toxicities are defined as side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment
Determine the recommended Phase 2 dose (RP2D) of MHB088C | through study completion, an average of 1 year
  The recommended phase 2 dose (RP2D) is determined traditionally by dose-limiting toxicities.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) parameter: Maximum concentration (Cmax) | Within 5 cycles (each cycle is 28 days)
  MHB088C, total antibody, free toxin MH30010008
PK parameter: Time to maximum concentration (Tmax) | Within 5 cycles (each cycle is 28 days)
  MHB088C, total antibody, free toxin MH30010008
PK parameter: Area under the concentration-time curve (AUC) | Within 5 cycles (each cycle is 28 days)
  MHB088C, total antibody, free toxin MH30010008
PK parameter: Trough concentration (Ctrough) | Within 5 cycles (each cycle is 28 days)
  MHB088C, total antibody, free toxin MH30010008
PK parameter: Terminal or apparent terminal half-life (t1/2) | Within 5 cycles (each cycle is 28 days)
  MHB088C, total antibody, free toxin MH30010008
PK parameter: Systemic clearance (CL) | Within 5 cycles (each cycle is 28 days)
  MHB088C, total antibody, free toxin MH30010008
Immunogenicity Assessment | Within 5 cycles (each cycle is 28 days)
  Assessment of anti-drug antibody (ADA)
Objective Response Rate (ORR) | through study completion, an average of 1 year
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR)
Duration of Response (DOR) | through study completion, an average of 1 year
  DOR was defined as the time from first assessment of PR or CR until disease progression.
Disease Control Rate (DCR) | through study completion, an average of 1 year
  DCR was defined as the proportion of participants with a complete response (CR), partial response (PR) or stable disease (SD).
Progression Free Survival (PFS) | through study completion, an average of 1 year
  Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Pindara Private Hospital, Gold Coast, Queensland
  - Southern Oncology Clinical Research Unit, Adelaide, South Australia
  - Cabrini Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Undecided